CLINICAL TRIAL: NCT04030598
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 2a Study to Assess the Clinical Efficacy of ISIS 721744, a Second-Generation Ligand-Conjugated Antisense Inhibitor of Prekallikrein, in Patients With Hereditary Angioedema
Brief Title: A Study to Assess the Clinical Efficacy of Donidalorsen (Also Known as IONIS-PKK-LRx and ISIS 721744) in Participants With Hereditary Angioedema
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ISIS 721744-CS2; 2019-001044-22 (EudraCT Number)
Record Dates: First submitted 2019-07-22; First posted 2019-07-24 (Actual); Results first posted 2022-09-28 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Hereditary Angioedema
Keywords: IONIS PKK-LRx; Donidalorsen
MeSH Terms: conditions — Angioedemas, Hereditary | interventions — donidalorsen; IONIS-PKK-LRx

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Part A was randomized, double-blind; Part B was open-label.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Part A: Placebo (Placebo Comparator): Participants with hereditary angioedema type I/type II (HAE-1/HAE-2) received placebo subcutaneously (SC) every 4 weeks at Weeks 1, 5, 9, and 13.
  Interventions: Drug: Placebo
- Part A: Donidalorsen 80 mg (Experimental): Participants with HAE-1/HAE-2 received donidalorsen, 80 mg, SC, every 4 weeks at Weeks 1, 5, 9, and 13.
  Interventions: Drug: Donidalorsen
- Part B: Donidalorsen 80 mg (Experimental): Participants with hereditary angioedema with normal C1-inhibitor (HAE-nC1-INH) received donidalorsen, 80 mg, SC, every 4 weeks at Weeks 1, 5, 9, and 13.
  Interventions: Drug: Donidalorsen

INTERVENTIONS:
Drug: Donidalorsen — Donidalorsen administered SC
  Other Names: ISIS 721744; IONIS-PKK-LRx
  Arms: Part A: Donidalorsen 80 mg; Part B: Donidalorsen 80 mg
Drug: Placebo — Placebo matching solution administered SC
  Arms: Part A: Placebo

SUMMARY:
The purpose of this study was to evaluate the clinical efficacy, safety, and tolerability of donidalorsen in participants with hereditary angioedema (HAE) type 1 (HAE-1), HAE type 2 (HAE-2), or HAE with normal C1-inhibitor (C1-INH) and to evaluate the effect of donidalorsen on plasma prekallikrein (PKK) and other relevant biomarkers.

DETAILED DESCRIPTION:
This was a randomized, double-blind, placebo-controlled study in 23 participants conducted concurrently in 2 parts (Part A and Part B); participants were allocated into Part A or Part B according to type of HAE (i.e., either HAE-1/HAE-2 in Part A or HAE-nC1-INH in Part B). Part A was randomized, double-blind, and placebo-controlled; and Part B was open-label. The length of participation in the study was approximately 8 months, which included an up to 8-week screening period, a 12-week treatment period, and a 13-week post-treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of HAE-1/HAE-2 (for inclusion in Part A) or HAE-nC1-INH (for inclusion in Part B)
* Participants must have experienced a minimum of 2 HAE attacks (assessed by the Angioedema Activity Score [AAS] and confirmed by the investigator) during the screening period
* Access to, and the ability to use, ≥ 1 acute medication(s) to treat angioedema attacks

Exclusion Criteria:

* Anticipated use of short-term prophylaxis for angioedema attacks for a pre-planned procedure during the screening or study periods
* Concurrent diagnosis of any other type of recurrent angioedema, including acquired or idiopathic angioedema
* Known history of or positive test for human immunodeficiency virus (HIV), hepatitis C, or chronic hepatitis B
* Malignancy within 5 years, except for basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix that has been successfully treated
* Treatment with another investigational drug or biological agent within 1 month or 5 half-lives, whichever is longer, of screening
* Exposure to any of the following medications:

  * Angiotensin-converting enzyme (ACE) inhibitors or any estrogen-containing medications with systemic absorption (such as oral contraceptive or hormonal replacement therapy) within 4 weeks prior to screening
  * Chronic prophylaxis with Lanadelumab within 10 weeks prior to screening
  * Oligonucleotides (including small interfering ribonucleic acid [RNA]) within 4 months of screening (if single dose received) or within 12 months of screening (if multiple doses received)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2020-01-07 (Actual); Primary Completion 2021-01-04 (Actual); Study Completion 2021-03-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (7):
  - Medical Research of Arizona, Scottsdale, Arizona
  - University of California San Diego (UCSD), San Diego, California
  - AIRE Medical of Los Angeles, Santa Monica, California
  - Midwest Immunology Clinical, Plymouth, Minnesota
  - Bernstein Clinical Research Center, LLC, Cincinnati, Ohio
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - AARA Research Center, Dallas, Texas
- Amsterdam UMC, loc. AMC, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fijen LM, Riedl MA, Bordone L, Bernstein JA, Raasch J, Tachdjian R, Craig T, Lumry WR, Manning ME, Alexander VJ, Newman KB, Revenko A, Baker BF, Nanavati C, MacLeod AR, Schneider E, Cohn DM. Inhibition of Prekallikrein for Hereditary Angioedema. N Engl J Med. 2022 Mar 17;386(11):1026-1033. doi: 10.1056/NEJMoa2109329. PMID 35294812

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 7 investigative sites from 7 January 2020 to 1 March 2021.
Pre-assignment Details: Participants with hereditary angioedema were concurrently enrolled in Part A and B, respectively. In Part A, 20 participants with hereditary angioedema type I/type II (HAE-1/HAE-2) were randomized in 2:1 ratio to receive donidalorsen or placebo for 13 weeks. In Part B, 3 participants with hereditary angioedema with normal C1-inhibitor (HAE-nC1-INH) received donidalorsen for 13 weeks after Part A.
Period: Overall Study
Arm/Group | Part A: Placebo | Part A: Donidalorsen 80 mg | Part B: Donidalorsen 80 mg
Started | 6 | 14 | 3
Completed (Completed=Participants who completed study treatment) | 6 | 13 | 3
Not Completed | 0 | 1 | 0
Not completed — Voluntary Withdrawal | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The safety population included all enrolled participants who received at least 1 dose of study drug (donidalorsen or placebo).
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A: Placebo | Part A: Donidalorsen 80 mg | Part B: Donidalorsen 80 mg | Total
Number analyzed (Participants) | 6 | 14 | 3 | 23
Age, Continuous [Mean (Full Range); unit: years] | 40.0 [22 to 56] | 37.8 [21 to 66] | 34.0 [25 to 40] | 37.26 [21 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 9 | 3 | 16
  Male | 2 | 5 | 0 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 6 | 13 | 3 | 22
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1
  White | 5 | 14 | 3 | 22
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Time-normalized Number of HAE Attacks (Per Month) From Week 1 to Week 17
Description: The Week 1 to end of on-treatment period HAE attack rate was calculated for each participant as number of HAE attacks occurring from Week 1 to 28 days after the last dose date divided by the number of days the participant contributed to the period multiplied by 28 days. An HAE attack was defined as an event with signs or symptoms consistent with an attack in at least 1 of the locations: peripheral angioedema (cutaneous swelling involving an extremity, the face, neck, torso, and/or genitourinary region), abdominal angioedema (abdominal pain, with or without abdominal distention, nausea, vomiting, or diarrhea), laryngeal angioedema (stridor, dyspnea, difficulty speaking, difficulty swallowing, throat tightening, or swelling of the tongue, palate, uvula, or larynx).
Time Frame: Week 1 to Week 17
Population: The intent-to-treat (ITT) population included all enrolled or randomized participants.
Measure: Mean (Standard Deviation); unit: HAE attacks per month
Groups:
- Part A: Placebo: Participants with HAE-1/HAE-2 received placebo subcutaneously (SC) every 4 weeks at Weeks 1, 5, 9, and 13.
Arm/Group | Part A: Placebo | Part A: Donidalorsen 80 mg | Part B: Donidalorsen 80 mg
Number analyzed (Participants) | 6 | 14 | 3
HAE attacks per month | 2.21 (1.558) | 0.23 (0.268) | 1.52 (2.221)
Statistical Analysis 1: Comparison: Part A: Placebo vs Part A: Donidalorsen 80 mg; Test type: Superiority; p = 0.001, Wald Chi-Square; Percentage Difference = -90.00, 95% CI 2-sided [-96.00 to -76.00] — The percentage difference in mean investigator-confirmed HAE attack rate between donidalorsen 80 mg and placebo was calculated as 100 percentage (%) × (mean rate ratio -1)

2. Secondary Outcome: Time-normalized Number of Investigator-confirmed HAE Attacks (Per Month) From Week 5 to Week 17
Description: The Week 5 to end of on-treatment period HAE attack rate was calculated for each participant as number of HAE attacks occurring from Week 5 to 28 days after the last dose date divided by the number of days the participant contributed to the period multiplied by 28 days. An HAE attack was defined as an event with signs or symptoms consistent with an attack in at least 1 of the locations: peripheral angioedema (cutaneous swelling involving an extremity, the face, neck, torso, and/or genitourinary region), abdominal angioedema (abdominal pain, with or without abdominal distention, nausea, vomiting, or diarrhea), laryngeal angioedema (stridor, dyspnea, difficulty speaking, difficulty swallowing, throat tightening, or swelling of the tongue, palate, uvula, or larynx).
Time Frame: Week 5 to Week 17
Population: ITT population included all enrolled or randomized participants.
Measure: Mean (Standard Deviation); unit: HAE attacks per month
Arm/Group | Part A: Placebo | Part A: Donidalorsen 80 mg | Part B: Donidalorsen 80 mg
Number analyzed (Participants) | 6 | 14 | 3
HAE attacks per month | 2.06 (1.574) | 0.07 (0.267) | 1.78 (2.795)
Statistical Analysis 1: Comparison: Part A: Placebo vs Part A: Donidalorsen 80 mg; Test type: Superiority; p = 0.003, Wald Chi-Square; Percentage Difference = -89.00, 95% CI 2-sided [-95.00 to -77.00] — The percentage difference in mean investigator-confirmed HAE attack rate between donidalorsen 80 mg and placebo was calculated as 100% × (mean rate ratio -1)

3. Secondary Outcome: Time-normalized Number of Moderate or Severe Investigator-confirmed HAE Attacks (Per Month) From Week 5 to Week 17
Description: The Week 5 to end of on-treatment period HAE attack rate was calculated for each participant as number of moderate or severe HAE attacks occurring from Week 5 to 28 days after the last dose date divided by the number of days the participant contributed to the period multiplied by 28 days. An HAE attack was defined as an event with signs or symptoms consistent with an attack in at least 1 of the locations: peripheral angioedema (cutaneous swelling involving an extremity, the face, neck, torso, and/or genitourinary region), abdominal angioedema (abdominal pain, with or without abdominal distention, nausea, vomiting, or diarrhea), laryngeal angioedema (stridor, dyspnea, difficulty speaking, difficulty swallowing, throat tightening, or swelling of the tongue, palate, uvula, or larynx). HAE attack severity: Mild: transient or mild discomfort, Moderate: mild to moderate limitation in activity, some assistance needed, and Severe: marked limitation in activity, assistance required.
Time Frame: Week 5 to Week 17
Population: ITT population included all enrolled or randomized participants.
Measure: Mean (Standard Deviation); unit: HAE attacks per month
Arm/Group | Part A: Placebo | Part A: Donidalorsen 80 mg | Part B: Donidalorsen 80 mg
Number analyzed (Participants) | 6 | 14 | 3
HAE attacks per month | 1.25 (1.208) | 0.05 (0.178) | 0.89 (1.540)
Statistical Analysis 1: Comparison: Part A: Placebo vs Part A: Donidalorsen 80 mg; Test type: Superiority; p = 0.004, Wald Chi-Square; Percentage Difference = -96.00, 95% CI 2-sided [-100.00 to -65.00] — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: Number of Participants With Clinical Response by Week 17
Description: Clinical response was defined as a ≥ 50%, ≥ 70%, or ≥ 90% reduction from Baseline in HAE attack rate from Week 5 to Week 17. The HAE attack rate was calculated as number of investigator-confirmed HAE attacks occurring from Week 5 to 28 days after last dose administration, divided by the number of days the participant contributed to the period multiplied by 28 days. An HAE attack was defined as an event with signs or symptoms consistent with an attack in at least 1 of the locations: peripheral angioedema (cutaneous swelling involving an extremity, the face, neck, torso, and/or genitourinary region), abdominal angioedema (abdominal pain, with or without abdominal distention, nausea, vomiting, or diarrhea), laryngeal angioedema (stridor, dyspnea, difficulty speaking, difficulty swallowing, throat tightening, or swelling of the tongue, palate, uvula, or larynx).
Time Frame: Week 5 to Week 17
Population: ITT population included all enrolled or randomized participants. Overall number of participants analyzed is the number of participants with data available for analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo | Part A: Donidalorsen 80 mg | Part B: Donidalorsen 80 mg
Number analyzed (Participants) | 6 | 13 | 3
Participants
  ≥ 50% Reduction | 2 | 13 | 2
  ≥ 70% Reduction | 1 | 12 | 2
  ≥ 90% Reduction | 0 | 12 | 1
Statistical Analysis 1: Comparison: Part A: Placebo vs Part A: Donidalorsen 80 mg; For ≥ 50% reduction from Baseline in the HAE attack rate; Test type: Superiority; p = 0.004, Fisher Exact; Risk Difference (RD) = 66.7, 95% CI 2-sided [17.5 to 95.7]
Statistical Analysis 2: Comparison: Part A: Placebo vs Part A: Donidalorsen 80 mg; For ≥ 70% reduction from Baseline in the HAE attack rate; Test type: Superiority; p = 0.003, Fisher Exact; Risk Difference (RD) = 75.6, 95% CI 2-sided [26.8 to 96.5]
Statistical Analysis 3: Comparison: Part A: Placebo vs Part A: Donidalorsen 80 mg; For ≥ 90% reduction from Baseline in the HAE attack rate; Test type: Superiority; p < 0.001, Fisher Exact; Risk Difference (RD) = 92.3, 95% CI 2-sided [48.0 to 99.8]

5. Secondary Outcome: Number of Investigator-confirmed HAE Attacks Requiring Acute Therapy From Week 5 to Week 17
Description: The Week 5 to end of on-treatment period HAE attack rate was calculated for each participant as number of HAE attacks requiring acute therapy occurring from Week 5 to 28 days after the last dose date divided by the number of days the participant contributed to the period multiplied by 28 days. An HAE attack was defined as an event with signs or symptoms consistent with an attack in at least 1 of the locations: peripheral angioedema (cutaneous swelling involving an extremity, the face, neck, torso, and/or genitourinary region), abdominal angioedema (abdominal pain, with or without abdominal distention, nausea, vomiting, or diarrhea), laryngeal angioedema (stridor, dyspnea, difficulty speaking, difficulty swallowing, throat tightening, or swelling of the tongue, palate, uvula, or larynx). HAE attacks requiring acute therapy included those attacks with medical intervention or hospitalization marked on the case report form (CRFs).
Time Frame: Week 5 to Week 17
Population: ITT population included all enrolled or randomized participants.
Measure: Mean (Standard Deviation); unit: HAE attacks per month
Arm/Group | Part A: Placebo | Part A: Donidalorsen 80 mg | Part B: Donidalorsen 80 mg
Number analyzed (Participants) | 6 | 14 | 3
HAE attacks per month | 1.25 (1.208) | 0.05 (0.178) | 0.89 (1.540)
Statistical Analysis 1: Comparison: Part A: Placebo vs Part A: Donidalorsen 80 mg; Test type: Superiority; p = 0.009, Wald Chi-Square; Percentage Difference = -95.00, 95% CI 2-sided [-99.00 to -52.00]

6. Secondary Outcome: Percentage of Cleaved High Molecular Weight Kininogen (cHMWK) Levels at Weeks 9 and 17
Description: High-molecular-weight kininogen (HMWK) is an abundant protein found in plasma and it has a critical role in acute attacks of HAE. During HAE attack plasma kallikrein cleaves HMWK producing cleaved HMWK (cHMWK) and bradykinin, the major biologic peptide that promotes the edema, one of the characteristic traits of HAE. Percentage of cHMWK levels were assessed to evaluate pharmacodynamics of donidalorsen.
Time Frame: Weeks 9 and 17
Population: ITT population included all enrolled or randomized participants. Number analyzed is number of participants with data available for analysis at specified time point.
Measure: Mean (Standard Deviation); unit: percentage of cHMWK levels
Arm/Group | Part A: Placebo | Part A: Donidalorsen 80 mg | Part B: Donidalorsen 80 mg
Number analyzed (Participants) | 6 | 14 | 3
percentage of cHMWK levels
  Week 9 | 5.62 (3.255) | 2.07 (1.241) | 1.03 (0.115)
  Week 17: number analyzed (Participants) | 6 | 13 | 3
  Week 17 | 7.00 (4.338) | 2.35 (1.353) | 2.13 (0.929)

7. Secondary Outcome: Prekallikrein (PKK) Activity Levels at Weeks 9 and 17
Description: Prekallikrein (PKK) has a critical role in acute attacks of HAE. During HAE attack PKK is activated to form plasma kallikrein. Plasma kallikrein cleaves HMWK producing cleaved HMWK (cHMWK) and bradykinin, the major biologic peptide that promotes the edema, one of the characteristic traits of HAE. Prekallikrein levels were measured to assess pharmacodynamics of donidalorsen.
Time Frame: Weeks 9 and 17
Population: ITT population included all enrolled or randomized participants. Number analyzed is number of participants with data available for analysis at specified timepoint.
Measure: Mean (Standard Deviation); unit: milligram per liter (mg/L)
Arm/Group | Part A: Placebo | Part A: Donidalorsen 80 mg | Part B: Donidalorsen 80 mg
Number analyzed (Participants) | 6 | 14 | 3
milligram per liter (mg/L)
  Week 9 | 95.467 (23.7193) | 37.676 (14.5639) | 25.630 (19.2671)
  Week 17: number analyzed (Participants) | 6 | 13 | 2
  Week 17 | 98.600 (34.5944) | 37.795 (38.6618) | 28.615 (22.8042)

8. Secondary Outcome: Number of Participants Who Consumed On-demand Medication at Weeks 9 and 17
Description: Treatment options for HAE included on-demand treatment of attacks and prophylaxis. On-demand medication options included supplementation of C1-INH (either plasma-derived or recombinant C1-INH concentrate) and inhibition of BK2 receptor activation (BK2-receptor antagonist). The number of participants who used on-demand medication at Week 9 (Day 57) and at Week 17 (end of the on-treatment period) were reported.
Time Frame: Weeks 9 and 17
Population: ITT population included all enrolled or randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo | Part A: Donidalorsen 80 mg | Part B: Donidalorsen 80 mg
Number analyzed (Participants) | 6 | 14 | 3
Participants
  Week 9 | 6 | 12 | 3
  Week 17 | 6 | 11 | 3
Statistical Analysis 1: Comparison: Part A: Placebo vs Part A: Donidalorsen 80 mg; Week 9; Test type: Superiority; p = 1.000, Fisher Exact; Risk Difference (RD) = -14.3, 95% CI 2-sided [-59.1 to 33.9]
Statistical Analysis 2: Comparison: Part A: Placebo vs Part A: Donidalorsen 80 mg; Week 17; Test type: Superiority; p = 0.521, Fisher Exact; Risk Difference (RD) = -21.4, 95% CI 2-sided [-64.9 to 27.1]

9. Secondary Outcome: Change From Baseline in Angioedema Quality of Life (AE-QoL) Questionnaire Total Score at Weeks 9 and 17
Description: The AE-QoL was developed to measure health-related quality of life (HRQoL) impairment in participants with recurrent angioedema. The AE-QoL is a self-administered questionnaire that can be completed in less than 5 minutes. It comprises 17 items across 4 domains: functioning, fatigue/mood, fears/shame, and food. Responses use a 5-point Likert scale ranging from '0 = never' to '4 = very often.' Per-participant scores for each domain were computed using the appropriate scoring algorithm applied to the question response scores for each domain. Per-participant total scores (including all 4 domains) were similarly computed using the question response scores for all 17 questions. The outputs from the scoring algorithm were normalized on a scale ranging from 0 (less adverse impact) to 100 (most adverse impact). Global total score ranges from 0 to 100, with higher scores indicating greater impairment. Mixed model for repeated measures (MMRM) was used for analyses.
Time Frame: Baseline, Weeks 9 and 17
Population: ITT population included all enrolled or randomized participants. Number analyzed is the number of participants with data available at specified timepoint.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Part A: Placebo | Part A: Donidalorsen 80 mg | Part B: Donidalorsen 80 mg
Number analyzed (Participants) | 6 | 14 | 3
score on a scale
  Change from Baseline at Week 9 | -1.50 (4.413) | -27.42 (2.854) | 25.49 (17.421)
  Change from Baseline at Week 17: number analyzed (Participants) | 6 | 13 | 3
  Change from Baseline at Week 17 | -6.15 (4.671) | -26.85 (3.133) | 26.96 (20.918)
Statistical Analysis 1: Comparison: Part A: Placebo vs Part A: Donidalorsen 80 mg; Week 9; Test type: Superiority; Treatment Difference = -25.92, 95% CI 2-sided [-37.10 to -14.74]
Statistical Analysis 2: Comparison: Part A: Placebo vs Part A: Donidalorsen 80 mg; Week 17; Test type: Superiority; Treatment Difference = -20.69, 95% CI 2-sided [-32.70 to -8.68]

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to end of the study (Up to Week 26)
Description: The safety population included all enrolled participants who received at least 1 dose of study drug (donidalorsen or placebo).
Arm/Group | Part A: Placebo | Part A: Donidalorsen 80 mg | Part B: Donidalorsen 80 mg
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/14 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/14 | 0/3
Other Adverse Events (participants affected / at risk) | 3/6 | 2/14 | 3/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Placebo (N=6) | Part A: Donidalorsen 80 mg (N=14) | Part B: Donidalorsen 80 mg (N=3)
Nausea (Gastrointestinal disorders) | 1 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 2 | 2 | 0
Application site rash (General disorders) | 0 | 0 | 1
Feeling hot (General disorders) | 0 | 0 | 1
Hyperhidrosis (General disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-05): https://cdn.clinicaltrials.gov/large-docs/98/NCT04030598/Prot_SAP_003.pdf